CLINICAL TRIAL: NCT04082819
Title: Determining the Accuracy of the HeartBeat Algorithm for Calculating Blood Pressure
Brief Title: MediBeat - HeartBeat Observation Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SE Health (Other)
Collaborators: Centre for Aging and Brain Health Innovation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: MCD307-007-1920
Record Dates: First submitted 2019-09-04; First posted 2019-09-09 (Actual); Results first posted 2020-04-01 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Low Blood Pressure; Blood Pressure; High Blood Pressure; Hypertension; Hypotension
MeSH Terms: conditions — Hypotension; Hypertension | interventions — Sphygmomanometers

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Low Blood Pressure (Other): Low blood pressure (systolic: 0-129, diastolic: 0-79)
  Interventions: Device: Contec CMS50EW; Device: Sphygmomanometer
- Medium Blood Pressure (Other): Medium blood pressure (systolic: 130-160, diastolic: 80-100)
  Interventions: Device: Contec CMS50EW; Device: Sphygmomanometer
- High Blood Pressure (Other): High blood pressure (systolic: 161 or higher, diastolic: 101 or higher)
  Interventions: Device: Contec CMS50EW; Device: Sphygmomanometer

INTERVENTIONS:
Device: Contec CMS50EW — Participants' blood pressure will be measured 3 times with the wearable finger pulse oximeter at their study visit.
Device: Sphygmomanometer — Participants' blood pressure will be measured 4 times manually with a blood pressure cuff at their study visit.

SUMMARY:
The goal of the study was to compare the current gold standard blood pressure instrument (a mercury-filled sphygmomanometer with cuff and stethoscope) with the new experimental algorithm developed by HeartBeat Technologies Ltd. To that end, participants were recruited from Markham, Ontario and participated in a series of alternating blood pressure measurements over a period of 45 minutes. Comparisons were made between manual measurements and device measurements to determine the quality of the device readings. Measurements were taken by trained nurses and staff were consistent across the study duration.

DETAILED DESCRIPTION:
The gold standard instrument for blood pressure measurement is a mercury-filled sphygmomanometer with cuff and stethoscope (Canadian Agency for Drugs and Technologies in Health; Canadian Electronic Library, 2012). However, such a device is not the most convenient for client self-monitoring or virtual (remote) care. Thus, there is a desire for an accurate, reliable alternative for the traditional mercury-containing sphygmomanometer.

HeartBeat Technologies Ltd. ("Heartbeat") has developed a novel approach to measuring blood pressure after an initial blood pressure reading using the conventional measurement method, supplemented by specific characteristics of a person (age, gender, height, weight, and heart rate), has established a "baseline measurement" for the person. The "novel approach" uses a finger pulse oximeter, the Contec CMS50EW device (Figure 1) (manufactured by Contec Medical Systems Co., Ltd., Shanghai, People's Republic of China). The finger pulse oximeter detects the changes in blood volume directly below the person's skin and indirectly measures oxygen saturation in the blood. The measurement is in the form of a photoplethysmogram (PPG) which is captured by the Contec oximeter and then, by Bluetooth technology, transmitted to a smartphone or tablet. A HeartBeat application, called MediBeat, on the smartphone or tablet then transmits the PPG to a server where a proprietary algorithm analyzes the baseline measurement for the person and the PPG to calculate the person's current blood pressure.

Heartbeat's intent is that the current blood pressure reading would then be made available to both the client and the health provider through separate web-based interfaces. Providers would be able to log onto the HeartBeat web-based application from anywhere to review and monitor the blood pressure of multiple clients, while clients can log onto the application to track their own measurements.

ELIGIBILITY:
Inclusion Criteria:

* adult over 25 years of age

Exclusion Criteria:

* those who have heart arrhythmias,
* atrial fibrillations or atrial flutters,
* an inaudible Korotkoff sound,
* wounds of the upper arms/wrists, missing fingers, and/or
* an arm circumference of more than 55 cm will be excluded

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2019-10-04 (Actual); Primary Completion 2019-11-22 (Actual); Study Completion 2019-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Holyoke, PhD, Principal Investigator — SE Health
Locations (1):
- SE Health, Markham, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Holyoke P, Yogaratnam K, Kalles E. Web-Based Smartphone Algorithm for Calculating Blood Pressure From Photoplethysmography Remotely in a General Adult Population: Validation Study. J Med Internet Res. 2021 Apr 23;23(4):e19187. doi: 10.2196/19187. PMID 33890856

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy participants who were 25 years old and worked in Markham were recruited. Only healthy subjects were included; those who were under 25, had heart arrhythmias, atrial fibrillations or atrial flutters, an inaudible Korotkoff sound, wounds of the upper arms/wrists, missing fingers, and/or an arm circumference of more than 55 cm were excluded.
Period: Overall Study
Arm/Group | Low Blood Pressure | Medium Blood Pressure | High Blood Pressure
Started | 37 | 54 | 3
Completed | 37 | 54 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Blood Pressure | Medium Blood Pressure | High Blood Pressure | Total
Number analyzed (Participants) | 37 | 54 | 3 | 94
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.1 (10.1) | 44.2 (10.6) | 48.0 (12.2) | 42.7 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 31 | 2 | 65
  Male | 5 | 23 | 1 | 29
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Difference Between Systolic Manual Sphygmomanometer and Finger Pulse Oximeter Readings
Description: Each device reading was compared to the manual blood pressure reading taken before (R1) and after it (R2). The degree of alignment for systolic blood pressure was calculated by taking the difference between the two scores (manual and device). The reading with the best alignment was used.
Time Frame: 45 - 60 minutes
Population: The overall participants analyzed indicate the number of individuals who matched the ranges listed in the description for low, medium or high blood pressure categories, where they had blood pressure ranges falling between the respective values indicated for the systolic pressure measured.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Low Blood Pressure: Systolic score between 90 - 120mmHg.
- Medium Blood Pressure: Systolic score between 130 - 160mmHg.
- High Blood Pressure: Systolic score greater than 161mmHg.
Arm/Group | Low Blood Pressure | Medium Blood Pressure | High Blood Pressure
Number analyzed (Participants) | 37 | 54 | 3
mmHg | 3 (6) | 3 (6) | 11 (10)

2. Primary Outcome: Difference Between Diastolic Manual and Device Blood Pressure Readings
Description: Each device reading was compared to the manual reading before (R1) and after (R2) it, to calculate the degree of alignment. The difference of the device and R1, and the device and R2 were taken. The smaller number was used for results reporting.
Time Frame: 45-60 minutes
Population: The overall participants analyzed indicate the number of individuals who matched the ranges listed in the description for low, medium or high blood pressure categories, where they had blood pressure ranges falling between the respective values indicated for the diastolic pressure measured.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Low Diastolic Blood Pressure: Diastolic score between 40-79mmHg.
- Medium Diastolic Blood Pressure: Diastolic score between 80-100mmHg.
- High Diastolic Blood Pressure: Diastolic score greater than 101mmHg.
Arm/Group | Low Diastolic Blood Pressure | Medium Diastolic Blood Pressure | High Diastolic Blood Pressure
Number analyzed (Participants) | 37 | 54 | 3
mmHg | 1 (4) | 0 (6) | 3 (4)

ADVERSE EVENTS:
Time Frame: For each participant, adverse event phenomena were monitored from the initial informed consent process and up to the remuneration process in the data gathering visit. This took approximately 45 minutes for each participant, during which they were continuously in the presence of trained medical professionals. Following this active assessment period, there was no follow-up conducted with participants, but participants were able to contact the research team with any concerns that may have arisen.
Description: Adverse events or risks (for all-cause mortality, serious, or non-serious) were monitored throughout study duration, however, none were observed across the 94 study participants.
Arm/Group | Low Blood Pressure | Medium Blood Pressure | High Blood Pressure
All-Cause Mortality (participants affected / at risk) | 0/94 | 0/94 | 0/94
Serious Adverse Events (participants affected / at risk) | 0/94 | 0/94 | 0/94
Other Adverse Events (participants affected / at risk) | 0/94 | 0/94 | 0/94

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-04): https://cdn.clinicaltrials.gov/large-docs/19/NCT04082819/Prot_SAP_000.pdf